CLINICAL TRIAL: NCT06916585
Title: A Phase II Clinical Trial to Evaluate the Safety and Efficacy of Injectable AS1501 in the Treatment of Acute-on-chronic Liver Failure (ACLF)
Brief Title: Chinese Phase II Trail of AS1501 in Acute-on-chronic Liver Failure (ACLF) Patients
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shenzhen Third People's Hospital (Other)
Collaborators: Guangzhou 8th People's Hospital (Other); Shenzhen Zhongke Amshenn Pharmaceutical Co., Ltd. (Other)
Responsible Party: Principal Investigator, Jun chen, PHD, Shenzhen Third People's Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AS1501-CTP-Ⅱ-01
Record Dates: First submitted 2025-03-31; First posted 2025-04-08 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Acute-On-Chronic Liver Failure
MeSH Terms: conditions — Acute-On-Chronic Liver Failure | interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 0.5mg/kg (Experimental)
  Interventions: Drug: AS1501 for injection
- 1.0mg/kg (Experimental)
  Interventions: Drug: AS1501 for injection

INTERVENTIONS:
Drug: AS1501 for injection — Single administration, after 20 days of elution, enter continuous administration, once a week for 4 consecutive weeks

SUMMARY:
**Document Name: This Trial is a Phase II Clinical Study.docx** **Document Content:**

* This trial is a Phase II clinical study, conducted in two stages:
* **Phase IIa:** A sentinel, single-arm design will be employed. A total of 12 early ACLF subjects are expected to be enrolled in the 0.5 mg/kg dose group. The first 2 subjects will serve as sentinels and be enrolled sequentially to receive a single intravenous dose. If no drug-related SAEs (Serious Adverse Events) occur in these 2 sentinel subjects within 2 weeks after the first dose, the remaining 10 subjects will be enrolled. Otherwise, the dose will be reduced for further exploration. After receiving a single intravenous dose, subjects will undergo a 20-day washout period. If no drug-related ≥Grade 3 AEs (Adverse Events) occur during this 20-day washout period, and safety/tolerability is jointly confirmed by the investigator and sponsor, the subject will enter the multiple-dose phase (once weekly [Day 21 as the first dose of multiple administration], for 4 consecutive weeks). If any drug-related ≥Grade 3 AE occurs, the dose will be reduced for further exploration, with the specific dose determined by the sponsor and investigator. If a subject drops out during the washout period after a single dose, additional subjects may be enrolled to ensure at least 12 subjects enter the multiple-dose phase.
* After all 12 early ACLF subjects in the 0.5 mg/kg dose group complete continuous dosing, the DMC (Data Monitoring Committee) will assess the safety of this dose group. If any of the following occur in the 0.5 mg/kg group, the DMC will discuss whether to proceed with dose escalation:

> 1) ≥1/3 of subjects experience drug-related Grade 3 SAEs; > 2) Any drug-related Grade 4 or higher SAEs.

* If the DMC determines that dose escalation criteria are met, an additional 12 early ACLF subjects will be enrolled to receive the 1 mg/kg dose group. The same enrollment rules as the 0.5 mg/kg group apply: the first 2 subjects are sentinels receiving a single intravenous dose. If no drug-related SAEs occur in these sentinels within 2 weeks post-dose, the remaining 10 subjects will be enrolled. Post-single-dose administration, subjects will undergo a 20-day washout period. If no drug-related ≥Grade 3 AEs occur during this period, and safety/tolerability is confirmed, subjects will enter the multiple-dose phase (once weekly [Day 21 as the first dose], for 4 consecutive weeks). Dropouts during the washout period may be replaced to ensure at least 12 subjects enter the multiple-dose phase.
* After completing the 0.5 mg/kg and 1 mg/kg dose exploration studies, the investigator and sponsor may determine the recommended dose for Phase IIb based on cumulative safety, efficacy, and potential PK/PD results. Additional dose groups or alternative administration frequencies may also be explored.
* **Phase IIb:** A randomized (1:1), double-blind, placebo-controlled design will be used. A total of 72 ACLF subjects are expected to receive either AS1501 at the appropriate dose/frequency or placebo to further evaluate the efficacy and safety of AS1501 injection. The specific design will be finalized based on Phase IIa results and agreed upon by the investigator and sponsor.

ELIGIBILITY:
Inclusion Criteria:

* The age range for signing the informed consent form is between 18 and 75 years old
* According to the "Diagnosis and Treatment Guidelines for Liver Failure (2018 Edition)" issued by the Liver Failure and Artificial Liver Group of the Infectious Diseases Branch of the Chinese Medical Association and the Severe Liver Disease and Artificial Liver Group of the Hepatology Branch of the Chinese Medical Association, it has been diagnosed with chronic acute liver failure, with specific indicators including:

  1. Patients with chronic liver disease (chronic hepatitis B, autoimmune hepatitis, drug-induced hepatitis, etc.) and the acute attack factor is drugs;
  2. Serum TBil ≥ 10 × ULN or average daily increase ≥ 17.1 μ mol/L;
  3. Meet any of the following three criteria: A has a tendency to bleed, PTA ≤ 40% (or INR ≥ 1.5); B combined with hepatic encephalopathy; C combined with hepatorenal syndrome or ascites.
* Screening was conducted in the early stage of liver failure and did not meet the criteria for liver transplantation;
* Early manifestations of liver failure:

Extreme fatigue, accompanied by severe gastrointestinal symptoms such as anorexia, vomiting, and bloating; ALT and/or AST continue to significantly increase, and jaundice progressively deepens (TBil>171 μ mol/L or daily increase>17.1 μ mol/L); There is a tendency for bleeding, with 30%<PTA ≤ 40% (or 1.5 ≤ INR<1.9); No complications or other extrahepatic organ failure.

* During the screening period, serum TRAIL levels increased and were ≥ 3 times higher than normal human TRAIL levels;
* Can understand the informed consent form, voluntarily participate and sign the informed consent form;
* Capable of completing experiments in accordance with the research protocol;
* The subjects (including partners) are willing to voluntarily adopt effective contraceptive measures within 6 months after the last administration of the investigational drug.

Exclusion Criteria:

* Patients with a history of allergies or severe allergies to protein drugs (CTCAE v5.0 score>grade 3);
* Patients who have completed liver transplantation or plan to undergo liver transplantation within one month.
* ACLF patients in the middle and late stages; Severe grade III ascites or refractory ascites accompanied by stage III-IV hepatic encephalopathy.
* Individuals who have received artificial liver treatment within one week prior to screening.
* Individuals with malignant tumors or a history of malignant tumors in the past; Patients with lung cancer, liver cancer, pancreatic cancer, gastrointestinal tract and other tumors were diagnosed by imaging (ultrasound, CT or MRI) and tumor markers (AFP, CEA, CA125 or CA199, etc.) during the screening period or within one month before the screening period.
* Individuals who have undergone gastroscopy or imaging (abdominal B-ultrasound, CT, or MRI) during the screening period or within one month prior to screening, and whose results indicate a risk of severe varicose veins with bleeding.
* Subjects with acute kidney injury (AKI) defined by KDIGO criteria: (1) Scr elevation ≥ 26.5 μ mol/L (0.3mg/dL, 1mg/dL=88.4 μ mol/L) within 48 hours; (2) Scr increases by 1.5 times or more than the baseline value within 7 days; (3) Decreased urine output (<0.5ml/kg/h) and lasting for more than 6 hours.
* There are the following laboratory test values or abnormal test values: a. Blood routine: platelet count (PLT)<75 × 109/L, hemoglobin (HGB)<80g/L; b. PT-INR>1.9 or PTA<30%; c. Left ventricular ejection fraction (LVEF)<50%; Blood creatinine>1.5 × ULN.
* Patients with severe respiratory dysfunction, difficulty breathing, or failure.
* Severe infections that cannot be controlled by concomitant medications, including infections of major organs such as the abdominal cavity, lungs, urinary tract, and skin.
* HIV positive individuals, or active tuberculosis or syphilis infected individuals.
* Individuals with a history of unstable ischemic heart disease, congestive heart failure, myocardial infarction, stroke, severe arrhythmia, etc.
* Subjects with uncontrolled severe hypertension or diabetes.
* Pregnant or lactating women, or those who test positive for pregnancy.
* Participants in clinical trials of other drugs or medical devices within 30 days prior to randomization or within five drug half lives.
* Having undergone trauma or major surgery (e.g. requiring general anesthesia) within 28 days prior to the first administration of the investigational drug. Note: Participants who plan to undergo surgical procedures under local anesthesia are eligible to participate in the study.
* Any serious underlying medical or mental condition (such as alcohol or drug abuse), dementia, or change in mental state; Or any issues that may impair the subject's ability to receive or tolerate planned treatment at the research center, understand informed consent, or issues that the researcher deems taboo to participate in the study or confound the evaluation or study results specified in the protocol.
* Researchers believe that other conditions are not suitable for participating in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2025-04-15 (Estimated); Primary Completion 2027-11-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
The incidence of adverse events (AE) and serious adverse events (SAE) | 42days

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Share trial data for 12 months after the end of the trial
URL: https://ngdc.cncb.ac.cn/gsub/

REFERENCES:
- [Background] 李兰娟,韩涛.肝衰竭诊治指南（2018年版）.实用肝脏病杂志, 2019, 22(2):8
- [Background] Arroyo V, Moreau R, Kamath PS, Jalan R, Gines P, Nevens F, Fernandez J, To U, Garcia-Tsao G, Schnabl B. Acute-on-chronic liver failure in cirrhosis. Nat Rev Dis Primers. 2016 Jun 9;2:16041. doi: 10.1038/nrdp.2016.41. PMID 27277335

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2025-03-03): https://cdn.clinicaltrials.gov/large-docs/85/NCT06916585/Prot_ICF_000.pdf